CLINICAL TRIAL: NCT01236222
Title: Health Effects of Commuter Cycling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Lars Østergaard, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Cycling
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Prevention
Keywords: commuter cycling; fitness; metabolic syndrome; children
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Control group (No Intervention)
- Cycling to school (Experimental)
  Interventions: Behavioral: Cycling to school

INTERVENTIONS:
Behavioral: Cycling to school — Regular cycling to school
  Arms: Cycling to school

SUMMARY:
The purpose of this study is to determine whether cycling to school is effective in the prevention of the metabolic syndrome.

DETAILED DESCRIPTION:
Physical activity plays a crucial role in relation to prevent a clustering of risk factors. In adults a lower all-cause mortality has been found in those cycling to work compared to inactive commuters. It thus seems possible that cycling to school will entail health beneficial effects for children.

ELIGIBILITY:
Inclusion Criteria:

* passive commuted to school last 6 months, own a bike

Exclusion Criteria:

* less than 2 km to school

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Fitness | Day 0, Day 120
  Difference in VO2max determined by use of a metabolic cart

SECONDARY OUTCOMES:
Metabolic syndrome | Day 0, Day 120
  Metabolic syndrome as defined by the international diabetes federation based upon: obesity(from age and gender adjusted BMI),TG,HDL,blood pressure,glucose (fasting)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern Denmark, Odense, Denmark, Denmark

REFERENCES:
- [Derived] Ostergaard L, Borrestad LA, Tarp J, Andersen LB. Bicycling to school improves the cardiometabolic risk factor profile: a randomised controlled trial. BMJ Open. 2012 Oct 31;2(6):e001307. doi: 10.1136/bmjopen-2012-001307. Print 2012. PMID 23117560